CLINICAL TRIAL: NCT00075517
Title: Phase II Study Of Gemcitabine And Docetaxel In Patients With Inoperable Stage IIIB Or IIIB or IV Non-Small Cell Lung Cancer
Brief Title: Gemcitabine and Docetaxel in Treating Patients With Inoperable Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000346806; FRE-GERCOR-DOCEGEM-B00-2; EU-20331
Record Dates: First submitted 2004-01-09; First posted 2004-01-12 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2007-07

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; large cell lung cancer; squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Docetaxel; Gemcitabine

INTERVENTIONS:
Drug: docetaxel
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and docetaxel, use different ways to stop tumor cells from dividing so they stop growing or die. Giving more than one drug may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with docetaxel works in treating patients with inoperable stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with inoperable stage IIIB or IV non-small cell lung cancer treated with gemcitabine and docetaxel.

Secondary

* Determine the progression-free and overall survival of patients treated with this regimen.
* Determine the tolerance profile of this regimen in these patients.
* Determine the quality of life of patients treated with this regimen.

OUTLINE: This is a nonrandomized, multicenter study.

Patients receive docetaxel IV over 1 hour and gemcitabine IV over 2 hours on day 1. Treatment repeats every 15 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, after courses 6 and 12, and then every 3 months thereafter.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 42 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer of 1 of the following histologic subtypes:

  * Epidermoid carcinoma
  * Large cell carcinoma
  * Adenocarcinoma
* Stage IIIB (T4, any N, M0 OR any T, N3, M0) OR Stage IV disease
* Inoperable disease
* Measurable disease

  * At least 1 unidimensionally measurable lesion at least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 to 75

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Platelet count at least 100,000/mm^3
* Absolute neutrophil count at least 2,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic

* Bilirubin no greater than normal
* Transaminases no greater than 1.5 times normal
* Alkaline phosphatase no greater than 2.5 times normal

Renal

* Creatinine no greater than 2.3 mg/dL

Cardiovascular

* No uncontrolled cardiac insufficiency

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 6 months after study therapy
* No uncontrolled infection
* No other prior malignancy except curatively treated basal cell skin cancer or carcinoma in situ of the cervix
* No grade 3 or 4 brain disorder
* No intolerance to polysorbate 80 or cortisones

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy, including taxanes or gemcitabine
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy to more than 20% of the bone marrow
* No prior radiotherapy for lung cancer
* At least 4 weeks since other prior radiotherapy and recovered

Surgery

* No prior surgery for lung cancer

Other

* More than 30 days since prior clinical trial participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-09

PRIMARY OUTCOMES:
Response rate

SECONDARY OUTCOMES:
Progression-free survival
Overall survival
Tolerability
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Terrioux, MD — Clinique de Docteur Terrioux
Locations (12):
- France (12):
  - Hopital Avicenne, Bobigny
  - Centre Jean Bernard, Le Mans
  - Hopital Perpetuel Secours, Levallois-Perret
  - Centre de Radiotherapie et Oncologie Saint-Faron, Mareuil-lès-Meaux
  - Clinique de Docteur Terrioux, Meaux
  - American Hospital of Paris, Neuilly-sur-Seine
  - Hopital Tenon, Paris
  - Clinique les Bleuets, Reims
  - Polyclinique De Courlancy, Reims
  - Centre Rene Huguenin, Saint-Cloud
  - Clinique Francois, Saint-Dizier
  - Hopital Paul Brousse, Villejuif